CLINICAL TRIAL: NCT00576992
Title: A Clinical Study of Demographics and Findings During Endoscopy in Patients With Abdominal Pain, Dyspepsia, GERD, and Associated Symptoms
Brief Title: Demographics and Findings of Upper Endoscopy Patients
Status: Terminated | Type: Observational
Why Stopped: Recruitment not being met
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Principal Investigator, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: PS0014
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Barrett Esophagus; Gastroesophageal Reflux
Keywords: Barrett's Esophagus; Demographics; Questionnaire; Heartburn
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GI observation: Patients presenting for an upper endoscopy procedure with gastrointestinal symptoms or complaints.

SUMMARY:
The purpose of this study is to evaluate the demographics, patients symptoms, and findings during endoscopy. Patients presenting for an endoscopy procedure to the KCVA GI endoscopy suite, will be asked to fill out questionnaires pertaining to their symptoms and indications for the procedure. This will be done before their procedure during the interview period preceding endoscopy. The patient's answers to this questionnaire will aid us in determining the prevalence of gastric and esophageal disease in patients presenting with the complaints of dyspepsia, GERD, or extraesophageal symptoms and to also determine whether the presence of any factors (hiatal hernia, NSAID use, age, race, gender, etc.) contribute to the above endoscopic diagnoses.

DETAILED DESCRIPTION:
Barrett's esophagus is a pre-malignant condition associated with adenocarcinoma of the lower esophagus, and is found in 10-15% of patients with Gastroesophageal Reflux Disease (GERD). In prospective studies of patients undergoing endoscopy for reflux symptoms, the prevalence of long segments of Barrett's Esophagus (3cm or greater) is reported to be 3% and that of short segment Barrett's Esophagus (less than 3cm), to be approximately 7-8%. Early diagnosis with surveillance is considered the optimal approach in patients with Barrett's, given the poor survival of advanced adenocarcinoma of the esophagus. However, classic symptoms of GERD may be diminished in some patients with Barrett's esophagus, possibly leading to a lower incidence of endoscopy with early diagnosis.

Extraesophageal manifestations of GERD include hoarseness, wheezing, and globus sensation. Dyspepsia is defined as pain or discomfort centered in the upper abdomen. Some reports have quantified the incidence of dyspepsia as occurring in up to 40% of adults over a six-month period. The differential diagnosis of dyspepsia includes gastric or duodenal ulcer, gastroesophageal reflux disease, gastric cancer, and non-ulcer dyspepsia. The incidence of peptic ulcer disease appears to be decreasing in our population, largely due to the lower prevalence of Helicobacter pylori infection among the population. Thus, esophageal lesions are responsible for an increasing number of dyspeptic patients.

Controversies exist as to the proper management of patients presenting with dyspepsia. Empiric acid-suppression therapy is often the first step in the management of dyspeptic patients. Many physicians have adopted a test-and-treat strategy for Helicobacter pylori infection. Finally, upper endoscopy may be performed. This test is considered the gold standard for the diagnosis of esophageal and gastroduodenal lesions. The initial evaluation of dyspeptic patients may be modified by other factors in their presentation, i.e. age greater than 50 or the presence of alarm symptoms (weight loss, dysphagia, evidence of gastrointestinal bleeding, anemia, or previous gastric surgery).

A distinction between the various causes of dyspepsia is important to establish in view of the significant differences in treatment strategies. Several previously reported studies have established a correlation between dyspepsia, with or without peptic ulcer disease, and erosive esophagitis. These studies were limited by a high degree of patient selection and narrow patient populations. Although the prevalence of erosive esophagitis and Barrett's Esophagus has been reported in patients with typical GERD symptoms, i.e. heartburn and regurgitation, the exact prevalence in patients with atypical symptoms of GERD (cough, asthma, wheezing, dysphagia), abdominal pain and dyspepsia is not readily known, especially in a VA population. Given that these esophageal diseases affect mainly older Caucasian males, studying the prevalence of these diseases in a VA population would be of extreme significance and importance.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the KCVA GI endoscopy unit with symptoms of reflux,upper abdominal pain, anemia (patients referred by their primary care physicians with a diagnosis of low hemoglobin (< 10 G/DL, and or dyspepsia

Exclusion Criteria:

* Weight loss (Weight loss of > 10% of their mean body weight over last 6 months)
* Dysphagia
* Gastrointestinal bleeding
* Gastrointestinal malignancy
* Recent EGD (in the past 5 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is a Veteran population presenting to a VA Hospital upper endoscopy unit
Sampling Method: Non-Probability Sample
Enrollment: 1177 (Actual)
Dates: Start 2003-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of gastric and esophageal disease in patients presenting with the complaints of dyspepsia, GERD, or extraesophageal symptoms | 1 year

SECONDARY OUTCOMES:
Determine whether the presence of any factors (hiatal hernia, NSAID use, age, race, gender, etc.) contribute to the above endoscopic diagnoses | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Department of Veterans Affairs Medical Center of Kansas City
Locations (1):
- Department of Veterans Affairs Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Background] Sonnenberg A, El-Serag HB. Clinical epidemiology and natural history of gastroesophageal reflux disease. Yale J Biol Med. 1999 Mar-Jun;72(2-3):81-92. PMID 10780569
- [Background] Winters C Jr, Spurling TJ, Chobanian SJ, Curtis DJ, Esposito RL, Hacker JF 3rd, Johnson DA, Cruess DF, Cotelingam JD, Gurney MS, et al. Barrett's esophagus. A prevalent, occult complication of gastroesophageal reflux disease. Gastroenterology. 1987 Jan;92(1):118-24. PMID 3781178
- [Background] Johnston MH, Hammond AS, Laskin W, Jones DM. The prevalence and clinical characteristics of short segments of specialized intestinal metaplasia in the distal esophagus on routine endoscopy. Am J Gastroenterol. 1996 Aug;91(8):1507-11. PMID 8759651
- [Background] Hirota WK, Loughney TM, Lazas DJ, Maydonovitch CL, Rholl V, Wong RK. Specialized intestinal metaplasia, dysplasia, and cancer of the esophagus and esophagogastric junction: prevalence and clinical data. Gastroenterology. 1999 Feb;116(2):277-85. doi: 10.1016/s0016-5085(99)70123-x. PMID 9922307
- [Background] Knill-Jones RP. Geographical differences in the prevalence of dyspepsia. Scand J Gastroenterol Suppl. 1991;182:17-24. doi: 10.3109/00365529109109532. PMID 1896825
- [Background] Jones R, Lydeard S. Dyspepsia in the community: a follow-up study. Br J Clin Pract. 1992 Summer;46(2):95-7. PMID 1457318
- [Background] Voutilainen M, Sipponen P, Mecklin JP, Juhola M, Farkkila M. Gastroesophageal reflux disease: prevalence, clinical, endoscopic and histopathological findings in 1,128 consecutive patients referred for endoscopy due to dyspeptic and reflux symptoms. Digestion. 2000;61(1):6-13. doi: 10.1159/000007730. PMID 10671769
- [Background] de Moraes-Filho JP, Zaterka S, Pinotti HW, Bettarello A. Esophagitis and duodenal ulcer. Digestion. 1974;11(5-6):338-46. doi: 10.1159/000197601. No abstract available. PMID 4463131
- [Background] de Moraes-Filho JP. Lack of specificity of the acid perfusion test in duodenal ulcer patients. Am J Dig Dis. 1974 Sep;19(9):785-90. doi: 10.1007/BF01071936. No abstract available. PMID 4852636
- [Background] Flook D, Stoddard CJ. Gastro-oesophageal reflux and oesophagitis before and after vagotomy for duodenal ulcer. Br J Surg. 1985 Oct;72(10):804-7. doi: 10.1002/bjs.1800721010. PMID 4041712
- [Background] Earlam RJ, Amerigo J, Kakavoulis T, Pollock DJ. Histological appearances of oesophagus, antrum and duodenum and their correlation with symptoms in patients with a duodenal ulcer. Gut. 1985 Jan;26(1):95-100. doi: 10.1136/gut.26.1.95. PMID 3965370
- [Background] Goldman MS Jr, Rasch JR, Wiltsie DS, Finkel M. The incidence of esophagitis in peptic ulcer disease. Am J Dig Dis. 1967 Oct;12(10):994-9. doi: 10.1007/BF02233258. No abstract available. PMID 6045993